CLINICAL TRIAL: NCT05142761
Title: Quantitative Tension in Posterior Component Separation for Abdominal Wall Reconstruction
Brief Title: Tension in Posterior Component Separation for Abdominal Wall Reconstruction
Status: Completed | Type: Observational
Sponsor: Michael Rosen (Other)
Responsible Party: Sponsor-Investigator, Michael Rosen, Professor of Surgery, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Other Study IDs: 21-1034
Record Dates: First submitted 2021-11-17; First posted 2021-12-03 (Actual); Last update posted 2023-03-30 (Actual); Status verified 2023-03

CONDITIONS: Ventral Incisional Hernia
Keywords: ventral hernia repair; tension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Posterior component separation: Patients undergoing posterior component separation

SUMMARY:
The purpose of this study is to measure the changes in tension after each release in a standard posterior component separation during abdominal wall reconstruction.

DETAILED DESCRIPTION:
Myofascial component separation techniques are purported to reduce tension in abdominal wall reconstruction, but few objective data exist regarding tension reduction with posterior component separation (PCS) techniques. PCS techniques include several unique steps: division of the posterior rectus sheath, division of the posterior lamella of the internal oblique aponeurosis, and transversus abdominis release. Each of these releases carries a certain amount of morbidity, including neurovascular injuries, posterior sheath breakdowns, and musculofascial disruptions resulting in lateral hernias, and thus should only be undertaken if necessary to achieve physiologic tension. More importantly, during a PCS, the surgeon must achieve posterior elements apposition in the midline to allow an adequate pocket to deploy the mesh and avoid breakdown and interstitial hernias and recurrences. Further, the anterior sheath should be reapproximated to complete a functional abdominal wall reconstruction. During each procedure, the surgeon must assess the tension on the posterior closure and decide whether further release is necessary to achieve a safe, durable repair of the posterior elements.

Demographic information, including patient age, gender, BMI, history of diabetes, chronic immunosuppression, smoking history, and history of prior ventral hernia repairs will be captured in the Abdominal Core Health Quality Collaborative (ACHQC), per the investigators' practice standard. Additional intraoperative information collected will be hernia size, extent of posterior component separation, mesh size and type, and location of mesh placement. The ACHQC is a hernia-specific, nationwide registry for quality improvement, featuring prospectively-collected, surgeon-entered data.

The aim of this study is to determine the changes in abdominal wall tension with progressive PCS in abdominal wall reconstruction. The investigators also aim to quantify the reduction in tension on both the anterior and posterior elements of a PCS.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for abdominal wall reconstruction
* Patients able to provide informed consent

Exclusion Criteria:

* Patients unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing abdominal wall reconstruction with posterior component separation.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2022-08-02 (Actual); Study Completion 2022-09-02 (Actual)

PRIMARY OUTCOMES:
Tension changes in posterior component separation | Tension measurements will be recorded immediately during surgery
  The tension required to bring the anterior and posterior elements of the abdominal wall to the midline after each step of the posterior component separation will be measured with a scale designed by Cleveland Clinic Mechanical Prototype machinists. The scale, hooked to a clamp on the edge of the abdominal wall, will measure tension in pounds.

SECONDARY OUTCOMES:
Wound Morbidity | 30 days after surgery
Readmission | 30 days after surgery
  Readmission to the hospital
Reoperation | 30 days after surgery
  Reoperation on abdominal wall reconstruction
Ileus | 30 days after surgery
  Number of Ileus events in study subjects
Pulmonary complications | 30 days after surgery
  Number of pulmonary complications in study subjects
Short term hernia recurrences | 30 days
  Recurrence of hernia following study procedures

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Rosen, M.D., Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Comprehensive Hernia Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No